CLINICAL TRIAL: NCT03213743
Title: Expression Profiling of microRNA Following Administration of Dexmedetomidine in Patients Undergoing Procedures
Brief Title: Expression Profiling of microRNA Following Administration of Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Jinqiao Qian, Professor, First Affiliated Hospital of Kunming Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1stKunmingMCQJQ
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- before dexmedetomidine (Other): We took blood samples before the administration of dexmedetomidine to determine exression level of microRNA in the subjects.
  Interventions: Drug: Dexmedetomidine Injection

INTERVENTIONS:
Drug: Dexmedetomidine Injection — Investigators gave the patients loading dose of dexmedetomidine for 10 minutes and maintaining dose of dexmedetomidine for 20 minutes. Investigators took blood samples before and after the administration of dexmedetomidine.
  Other Names: Dex group

SUMMARY:
The purpose of the study is to find out the differential expression profiling of microRNA before and after adiministration of dexmedetomidine in patients undergoing procedures, and then investigators will do some in vitro studies to validate the functions of the microRNA.

DETAILED DESCRIPTION:
Background and objective: The use of dexmedetomidine may have benefits on the clinical outcomes of cardiac surgery. MicroRNAs are non-coding RNA sequences that act as regulators of gene expression. Investigators conduct a study to determine the role of microRNAs in cardioprotection mediated by dexmedetomidine.

Methods: In this study 3 patients were selected. The blood sample were taken before administration of dexmedetomidine.Investigators infused loading dose of dexmedetomidine for 10 minutes and maintaining dese of dexmedetomidine for 20 minutes.Thirty minutes after the administration, another blood samples were taken and stored in the liquid nitrogen and both the samples were marked. Those sample were analyzed for differentially expressed microRNA with Exiqon miRNA Array.

ELIGIBILITY:
Inclusion Criteria:

* The patients without arrithmia will undergo procedure.

Exclusion Criteria:

* The patients have bradycardia (hear rate is less than 60 beats per minute) or conduction block.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
microRNA differential expression | 30 minutes
  microRNA differential expression exerts cardioprotection effect on patients undergoing procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Jinqiao Qian, Ph.D, Principal Investigator — First Affiliated Hospital of Kunming Medical University
Locations (1):
- Jinqiao Qian, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No